CLINICAL TRIAL: NCT01886521
Title: Use of Lumbar Drain Versus Ventricular Drain to Remove Clots in Patients Admitted to the Neuro-ICU After Subarachnoid Hemorrhage (a Randomized Trial).
Brief Title: Use of Lumbar Drain to Remove Clots in Patients Admitted to the Neuro-ICU After Subarachnoid Hemorrhage.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Peter Birkeland, Staff surgeon, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37238
Record Dates: First submitted 2013-06-09; First posted 2013-06-26 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Subarachnoid Hemorrhage.
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar drain group (Experimental): Lumbar drain
  Interventions: Procedure: Lumbar drain
- Ventricular drain (Active Comparator): Ventricular drain
  Interventions: Procedure: Ventricular drain

INTERVENTIONS:
Procedure: Lumbar drain
  Arms: Lumbar drain group
Procedure: Ventricular drain
  Arms: Ventricular drain

SUMMARY:
Recently, a clinical trial showed that the use of lumbar drains compared to ventricular drain in patients suffering from subarachnoid hemorrhage resulted in less delayed ischemic neurological deficits but failed to show a clinical benefit after 6 months. The underlying assumption was, that the cerebrospinal fluid (CSF) obtained from lumbar drains has a higher concentration of blood than CSF from lumbar drains. The investigators decided to test this assumption. In this study, the investigators will randomize patients to either placement of a ventricular or a lumbar drain and analyze the CSF drainage on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the neuro-ICU with aneurysmal subarachnoid hemorrhage
* In need for CSF drainage based on clinical judgment

Exclusion Criteria:

* intraventricular clots
* intraparenchymal clots causing midline shift
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Accumulated Hb and bilirubin in CSF drainage | From drain placement to removal, in average 10 days.

SECONDARY OUTCOMES:
placement of a ventriculoperitoneal shunt | participants will be followed for the duration of hospital stay, in average 3 weeks
Lindegaard ratio (TCD) > 3 | the participants will be followed for the duration of hospital stay, in average 3 weeks
clinical signs of vasospasms | The participants will be followedd for the duration of hospital stay, in average 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Birkeland, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Neurosurgery, Odense University Hospital, Odense, Denmark